CLINICAL TRIAL: NCT07391709
Title: Investigation of the Protective Effect of Alpha Lipoic Acid on Ischemic Reperfusion Damage in Ischemic Priapism in Rats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trabzon Kanuni Education and Research Hospital (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, İbrahim Sibal, doctor, Trabzon Kanuni Education and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/2
Record Dates: First submitted 2026-01-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Priapism; Reperfusion Injury
Keywords: Priapism; Alpha Lipoic Acid; Ischemia-Reperfusion Injury; Antioxidant; Rat
MeSH Terms: conditions — Priapism; Reperfusion Injury | interventions — Reperfusion; Thioctic Acid

STUDY DESIGN:
Intervention Model Description: Randomised controlled group animal experiment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Healthy rats with no induction of ischemic priapism or reperfusion. No pharmacological treatment was administered.
- Ischemic priapism + reperfusion (Experimental): Ischemic priapism was induced by applying a tourniquet to the base of the penis for 4 hours, followed by reperfusion. No antioxidant or pharmacological treatment was given.
  Interventions: Procedure: Ischemic priapism + reperfusion
- Ischemic priapism + reperfusion + ALA (Experimental): Ischemic priapism was induced by a 4-hour penile base tourniquet followed by reperfusion. Alpha-lipoic acid (ALA) was administered intraperitoneally at a dose of 100 mg/kg, 30 minutes before reperfusion.
  Interventions: Procedure: Ischemic priapism + reperfusion + ALA; Drug: Ischemic priapism + reperfusion + ALA

INTERVENTIONS:
Procedure: Ischemic priapism + reperfusion — Ischemic priapism was induced by applying a tourniquet to the base of the penis for 4 hours, followed by reperfusion.
  Other Names: Penile ischemia-reperfusion injury model; Penile tourniquet-induced ischemic priapism; Experimental ischemic priapism model
  Arms: Ischemic priapism + reperfusion
Procedure: Ischemic priapism + reperfusion + ALA — Ischemic priapism was induced by applying a tourniquet to the base of the penis for 4 hours, followed by reperfusion.
  Other Names: Penile tourniquet-induced ischemic priapism; Experimental ischemic priapism model; Penile ischemia-reperfusion injury model
  Arms: Ischemic priapism + reperfusion + ALA
Drug: Ischemic priapism + reperfusion + ALA — Alpha-lipoic acid was administered intraperitoneally at a dose of 100 mg/kg, 30 minutes before reperfusion.
  Other Names: ALA; α-Lipoic acid
  Arms: Ischemic priapism + reperfusion + ALA

SUMMARY:
The condition known in medical terminology as 'Priapism' refers to the state of erection in the male sexual organ persisting partially or completely for more than 4 hours without sexual stimulation or orgasm. This 'prolonged and painful erection' is generally observed in young adults, although it can occur in all age groups, including the neonatal period. There are three main types: ischaemic (restricted blood flow), non-ischaemic (unrestricted blood flow), and recurrent 'prolonged and painful erection'. This disorder is believed to develop as a result of malfunctions in the mechanism that causes the male sexual organ to lose its erection (detumescence of the penis). Although the return of blood flow (reperfusion) to the tissue following the termination of 'long and painful erection' is necessary to preserve this structure that has been deprived of blood for a period of time, the return of blood flow itself initiates a mechanistic process that causes damage due to restricted blood flow and the return of blood flow to the tissue.

Currently, there is no effective and safe medical treatment used to prevent tissue damage caused by ischaemia-reperfusion injury in the treatment of 'long and painful erection'. Currently, there is no effective and safe medical treatment used in the treatment of 'long and painful erection' to prevent tissue damage resulting from ischaemia-reperfusion injury. Alpha-lipoic acid is an antioxidant found in some foods and naturally produced in the body. In this study, a model of 'long and painful erection' will be created in a total of 18 rats divided into 6 groups, and the possible biochemical and histopathological protective effects of alpha-lipoic acid against this condition will be investigated.

DETAILED DESCRIPTION:
Priapism refers to a prolonged erection lasting more than four hours without any sexual stimulation, caused by a dysfunction of the mechanisms that regulate penile swelling, rigidity, and relaxation . Pathophysiologically, there are three main types of priapism: ischaemic, non-ischaemic, and recurrent (stuttering). Ischemic (veno-occlusive, low-flow) priapism is the most common type. Sickle cell anaemia, vasoactive drug use, haematological dyscrasias, heparin therapy, haemodialysis, malignancies (local or metastatic), hyperlipidaemia parenteral nutrition therapy, and trauma are among the many conditions that can cause priapism. Acute ischaemic priapism represents a medical emergency and may subsequently lead to erectile dysfunction (ED) . Ischemia-reperfusion (I/R) injury occurs with the resolution of priapism. Although reperfusion is a necessary mechanism for the preservation of ischaemic tissue, reperfusion itself initiates a pathophysiological process that causes injury. With I/R injury, neutrophils, inflammatory cytokines, and adhesion molecules with increased thrombogenicity are activated, and free oxygen radicals develop with massive intracellular Ca release . Oxidative stress damages the cell membrane and has harmful effects on the tissue, leading to permanent cellular injury. Alpha-lipoic acid (ALA) is an 8-carbon molecule first isolated from bovine liver in 1950 that can cross the blood-brain barrier. It may also be referred to as 1,2-dithiolane-3-pentanoic acid or thioctic acid . Alpha-lipoic acid (ALA) is a natural substance found in certain foods and also synthesised in the body. It is abundant in animal and plant tissues rich in mitochondrial complexes. Among plants, spinach, broccoli, and tomatoes contain the highest amounts of lipoic acid. In animal tissues, it is most abundant in the kidneys, heart, and liver. ALA is an enzymatic cofactor involved in glucose and lipid metabolism and regulates gene transcription. ALA also acts as an antioxidant because it not only improves internal antioxidant systems but also restores them and supports their production or cellular accessibility. It also effectively removes heavy metals responsible for oxidative stress from the bloodstream. ALA's most unique feature compared to other antioxidants is that it reacts as both a lipid and water-soluble compound . Pharmacologically, ALA improves glycaemic control and diabetes mellitus-related polyneuropathies; it also effectively reduces toxicities associated with heavy metal poisoning. As an antioxidant, ALA directly eliminates free radicals, chelates transition metal ions, increases cytosolic glutathione and vitamin C levels, and prevents toxicities associated with their depletion . It is used in preclinical studies and clinically in AIDS, renal lithiasis, ethanol intoxication, cerebral ischaemia, stroke, Parkinson's disease, skin inflammation, diabetic neuropathy, radiation damage, and cataract disease . This study will examine the efficacy of ALA in alleviating reperfusion injury in rat models of ischaemic priapism using biochemical and histopathological methods.

Literature review:

Publications on the subject published in PubMed, ClinicalKey, EAU, AUA Guide, National Thesis Centre, and Google Scholar were reviewed. Publications on ischaemic priapism within priapism were reviewed. These publications included a detailed examination of the pathophysiology, aetiology, interventions and treatments of priapism, and experimentally induced ischaemic priapism models. Publications containing biochemical properties related to alpha-lipoic acid and experimental studies used for treatment purposes were examined. Publications containing biomarker and histopathological examinations of serum and tissue samples examined in animal experimental models with induced ischaemia-reperfusion were reviewed.

Objective: The aim of this experimental study is to investigate the possible effects of alpha-lipoic acid on this condition biochemically and histopathologically by creating a 'long and painful erection' model in rats.

ELIGIBILITY:
Inclusion Criteria:

• Adult male Sprague-Dawley rats weighing 350-400 g.

Exclusion Criteria:

* Animals with congenital anomalies, active infection, or systemic disease.
* Animals that died before completion of the experimental protocol.

Ages: 10 Weeks to 16 Weeks | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in serum total antioxidant status (TAS) measured by Erel spectrophotometric assay | 7 days after reperfusion
  Serum total antioxidant status (TAS) will be measured using the Erel spectrophotometric assay.Unit of Measure mmol Trolox equivalent/L
Change in serum total oxidant status (TOS) measured by Erel spectrophotometric assay | 7 days after reperfusion
  Serum total oxidant status (TOS) will be measured using the Erel spectrophotometric assay.Unit of Measure µmol H₂O₂ equivalent/L
Change in serum glutathione peroxidase (GPx) activity measured by spectrophotometric enzyme activity assay | 7 days after reperfusion
  Serum glutathione peroxidase (GPx) activity will be measured using a spectrophotometric enzyme activity assay.Unit of Measure U/L
Change in serum malondialdehyde (MDA) concentration measured by ELISA | 7 days after reperfusion
  Serum malondialdehyde (MDA) concentration will be measured using a commercial ELISA kit.Unit of Measure ng/mL
Change in serum ischemia-modified albumin (IMA) concentration measured by ELISA | 7 days after reperfusion
  Serum ischemia-modified albumin (IMA) concentration will be measured using a commercial ELISA kit.Unit of Measure U/mL

SECONDARY OUTCOMES:
Change in serum tumor necrosis factor-alpha (TNF-α) concentration measured by ELISA | 7 days after reperfusion
  Serum tumor necrosis factor-alpha (TNF-α) concentration will be measured using a commercial ELISA kit.Unit of Measure pg/mL
Change in penile tissue tumor necrosis factor-alpha (TNF-α) concentration measured by ELISA | 7 days after reperfusion
  Penile tissue tumor necrosis factor-alpha (TNF-α) concentration will be measured using a commercial ELISA kit and normalized to tissue protein content.Unit of Measure pg/mg protein

OTHER OUTCOMES:
Change in GRP78 protein expression in penile tissue measured by immunohistochemistry | 7 days after reperfusion
  GRP78 protein expression in penile tissue will be assessed using immunohistochemical semi-quantitative scoring.Unit of Measure Semi-quantitative score
Change in CHOP protein expression in penile tissue measured by immunohistochemistry | 7 days after reperfusion
  CHOP protein expression in penile tissue will be assessed using immunohistochemical semi-quantitative scoring.Unit of Measure Semi-quantitative score

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Experimental Animal Research Center, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No